CLINICAL TRIAL: NCT00550264
Title: Physician Awareness of and Communication About Hospital Readmissions
Brief Title: Study of Physician Awareness of and Communication About Patient Readmissions to the Hospital
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Harvard Risk Management Foundation (Other)
Responsible Party: Christopher L. Roy, MD, Brigham & Women's Hospital
Allocation: Randomized | Model: Single Group | Masking: None
Other Study IDs: 2006P001975; BWH
Record Dates: First submitted 2007-10-25; First posted 2007-10-29 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2011-06

CONDITIONS: Hospital Readmission
Keywords: Hospital Readmission; Continuity of Care; Quality of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Other: Automatic notification of readmissions
- 2 (No Intervention)

INTERVENTIONS:
Other: Automatic notification of readmissions — The experimental group physicians will receive automatic e-mail notification when a patient is readmitted, including contact information for the readmitting team.
  Arms: 1

SUMMARY:
Patients admitted to inpatient medicine services often require early hospital readmission, and often they are readmitted to different physician or team, potentially without the knowledge of the prior physician or team. Thus, physicians may lose the opportunity to share valuable information about readmitted patients, which may be detrimental to continuity of care and patient safety. The purpose of this study is to determine baseline awareness and communication rates among physicians regarding readmissions, and then measure the effect of automatic notification on these rates.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to the general medicine service at two academic medical centers, and unexpectedly readmitted within 14 days.

Exclusion Criteria:

* Patients readmitted to the same physician(s), or those whose readmission was planned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2007-02; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Physician Awareness and Communication Rates | Within 24 hours of readmission time

CONTACTS AND LOCATIONS:
Overall Officials: Christopher L Roy, MD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Brigham & Women's Hospital, Boston, Massachusetts, United States

REFERENCES:
- [Background] Roy CL, Kachalia A, Woolf S, Burdick E, Karson A, Gandhi TK. Hospital readmissions: physician awareness and communication practices. J Gen Intern Med. 2009 Mar;24(3):374-80. doi: 10.1007/s11606-008-0848-x. Epub 2008 Nov 4. PMID 18982395